CLINICAL TRIAL: NCT06148727
Title: Evaluation of Masticatory Performance and Patient Satisfaction for Conventional and 3D Printed Implant Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A20011122
Record Dates: First submitted 2023-08-16; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Each patient received two prostheses; conventional and 3D-printed implant overdentures. The succession of complete denture insertion was randomized to diminish the effect of the order of complete denture use on the results. First, each denture was used for three months, followed by two weeks of rest; then, the other denture type was delivered to the patient and used for another three months.
Who Masked: Investigator
Masking Description: The succession of complete denture insertion was randomized to diminish the effect of the order of complete denture use on the results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional heat cured overdenture group (Active Comparator): patients received 4 interforamenal implants connected by 3 bar assembly and conventional heat cured overdenture (Control Group)
  Interventions: Device: Dental implant placement; Device: Bar attachment
- 3d- printed overdenture group (Active Comparator): patients received 4 interforamenal implants connected by 3 bar assembly and 3d printed overdenture (Study Group)
  Interventions: Device: Dental implant placement; Device: Bar attachment

INTERVENTIONS:
Device: Dental implant placement — Procedure/ surgery: Surgical placement of dental implants, four interforaminal dental implants were placed
Device: Bar attachment — Device: attachment, implants were connected to each others by 3 implant assembly in a trapezoidal design implants were loaded after 3 months of osseo-integration Control Group: patients received coventionally constructed heat cured overdenture Study Group: patients received 3d printed overdenture

SUMMARY:
The aim of this crossover clinical study was the evaluation and comparison of masticatory performance and patient satisfaction for patients rehabilitated with conventional heat cured acrylic resin and 3D printed mandibular implant overdentures retained with bar attachment.

it was concluded that 3D printed implant overdenture showed promising results regarding chewing efficiency and patient satisfaction compared to conventionally fabricated implant overdenture.

DETAILED DESCRIPTION:
The aim of this crossover clinical study was the evaluation and comparison of masticatory performance and patient satisfaction for patients rehabilitated with conventional heat cured acrylic resin and 3D printed mandibular implant overdentures retained with bar attachment.

Materials and Methods: Twelve completely edentulous healthy participants received new conventional dentures. Four interforaminal implants were inserted in the mandible. After osseointegration, bar was constructed with trapezoidal configuration. Each patient received randomly the following overdentures using a crossover design: conventional heat cured acrylic resin overdenture, 3d printed overdenture ( developed by scanning of mandibular conventional overdenture). Masticatory performance was evaluated with the two-colour mixing ability test after 5, 10, 20, 30, and 50 masticatory cycles. Patient satisfaction was also measured using McGill Denture Satisfaction Questionnaire. Evaluation was done after 3 months of using each overdenture.

Conclusion: Within this clinical study limitations, 3D printed implant overdenture showed promising results regarding chewing efficiency and patient satisfaction compared to conventionally fabricated implant overdenture.

ELIGIBILITY:
Inclusion Criteria:

* adequate bone quantity [classes 1-3 according to [Lekholm and Zarb] of the mandible in the lateral incisor and first premolar regions to receive 4 implants
* adequate restorative space [12-15 mm from the mucosa of the mandibular ridge to the occlusal plane- Class I according to Ahuja and Cagna 23 for bar supported implant overdenture. This was verified by direct measurement of old denture
* Angel's class I maxillo-mandibular relationship.

Exclusion Criteria:

* include systemic diseases that contraindicate implant placement
* irradiation of the head and neck region
* chemotherapy within the past 3 years
* bone metabolic diseases as uncontrolled diabetes mellitus
* smoking habit

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Chewing efficiency | at time of insertion of prosthesis T(0), 3 months after insertion T(3).
  Chewing efficiency was assessed using the previously documented two-color mixing ability test (colorimetric method) as follow: Two samples were prepared from two colored chewing gums. Patients were asked to keep the gum sample intraorally for one minute then start to chew it for 5, 10, 20, 30 and 50 strokes respectively. Five samples were used for the tests, the samples were spat into clear plastic bags. All samples were evaluated after flattening to wafers of 1 mm thickness. scanned by Digital scanner from both sides stored in Adobe Photoshop® format (psd). Then the color range tool and histogram function were used to pick out the unmixed white parts of the image. Then the ratio of Unmixed Fraction (UF) was computed using the following formula: (Pixels white side a + Pixels white side b) - 2× Pixels of scale / 2 × Pixels all. As a reference scale, a scanned piece of unmixed gum was copied in each image
Patient satisfaction | at time of insertion of prosthesis T(0), 3 months after insertion T(3).
  The eight core of McGill Denture Satisfaction Questionnaire (MDSQ) items were used to record patient satisfaction with their mandibular complete removable denture. One question concerns overall satisfaction with existing prostheses, whereas the other seven questions refer to specific aspects that may influence overall satisfaction: ease of cleaning; ability to speak; comfort; aesthetics/appearance; and denture stability; chewing ability; chewing function. Respondents provided answers on a 100-mm visual analogue scale. Patients were encouraged to respond to the survey questionnaire after functioning with each type of denture for 3-months.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shady, MD, Principal Investigator — Mansoura University Faculty of Dentistry, Prosthodontics department
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nabil MS, Mahanna FF, Said MM. Evaluation of masticatory performance and patient satisfaction for conventional and 3D-printed implant overdentures: a randomized crossover study. BMC Oral Health. 2024 Jun 8;24(1):672. doi: 10.1186/s12903-024-04389-1. PMID 38851676